CLINICAL TRIAL: NCT00272207
Title: A Randomized Double-blinded Placebo Controlled Trial Assessing the Effect of the Oral Cannabinoid Nabilone on Pain and Quality of Life in Patients With Fibromyalgia
Brief Title: A Trial Assessing the Effect of Nabilone on Pain and Quality of Life in Patients With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Winnipeg Regional Health Authority (Other)
Collaborators: Valeant Canada Limited (Industry)
Responsible Party: Principal Investigator, Dr. Lena Galimova, MD, FRCPC, Winnipeg Regional Health Authority
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WPG2005#1974
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Cannabinoids; Nabilone; Cesamet; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nabilone — Oral nabilone, 0.5 mg x7 days, increased to 0.5 mg t.i.d x 2 weeks if patient tolerates, then increase if patient tolerating to 0.5 in am and 1.0 mg at hs x 1 week, then if patient tolerating, increase to 1.0 mg b.i.d x 1 week.
  Other Names: Cesamet

SUMMARY:
The purpose of the study is to determine whether or not the drug Nabilone significantly reduces pain and improves quality of life in patients with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a disease of unknown cause. People with fibromyalgia experience diffuse body pain, fatigue, sleep disturbance, and a generalized stiffness and swollen feeling. Fibromyalgia affects 2-6% of the general population, affecting females more commonly than males. Symptoms usually start between 20 and 55 years of age.

No medical treatment has been specifically approved for the management of fibromyalgia, however, there is strong evidence that some antidepressants, exercise, and patient education are effective in reducing the pain experienced by fibromyalgia patients. A recent study of four patients has suggested the possible benefit of Nabilone, a synthetic cannabinoid, in the treatment of fibromyalgia, however more studies are needed.

Marijuana is the common name for cannabis. Nabilone (brand name, CESAMET®), is a synthetic cannabinoid (form of cannabis). Cannabinoid receptors exist naturally in the human body and respond to naturally occurring cannabinoids produced by the body, as well as marijuana and synthetic cannabinoids like Nabilone.

In Canada, Nabilone is approved for the treatment and management of severe nausea and vomiting associated with cancer chemotherapy and may be prescribed by physicians.

Research has shown that activating the cannabinoid receptors also has an effect on reducing acute and chronic pain.

Our hypothesis is that the synthetic cannabinoid Nabilone will significantly reduce the pain experienced by patients with fibromyalgia and improve quality of life, compared to the placebo controlled group. This will be evident by finding significant differences in Visual Analogue Scale pain scores, number of tender points, average pain threshold, and scores on the Fibromyalgia Impact Questionaire.

ELIGIBILITY:
Inclusion Criteria:

* The patient meets The American College of Rheumatology (1990) criteria for the classification of fibromyalgia. [5]
* 18-70 years old.
* Any gender.
* The patient has not received benefit from a tricyclic antidepressant, muscle relaxant, acetaminophen or non-steroidal anti-inflammatories for management of their pain.
* No previous use of oral cannabinoids for pain management.

Exclusion Criteria:

* The patient's pain is better explained by a diagnosis other then fibromyalgia.
* Abnormalities on routine baseline blood work including electrolytes, urea and creatinine, a complete blood count, and liver function tests (AST ALT GGT, Alk Phos, and LDH). Normal tests taken within 3 months prior to the study will be accepted if there is no history of acute illness since the time the blood was drawn.
* Heart disease. (Cannabinoids can reduce heart rate and blood pressure) Patients with heart disease will be excluded based on a history of angina, MI or CHF as well as a clinical exam.
* Schizophrenia or other Psychotic disorder
* Severe liver dysfunction. (Patients will be excluded if there is an elevation of any of the baseline liver enzymes)
* History of untreated non-psychotic emotional disorders.
* Cognitive impairment.
* Major illness in another body area.
* Pregnancy.
* Nursing mothers.
* Patients less than 18 years old.
* History of drug dependency.
* A known sensitivity to marijuana or other cannabinoid agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale Pain Scores | Baseline, then at week 2, 4 and 8
  Patient is asked to mark their pain from 0 to 10, with 0 = no pain, and 10 = worst pain imaginable
Number of Tender Points | At baseline, then at the week 2, 4 and 8 visits
  Physician examines by digital palpation for pain at each of the 18 characteristic tender points for fibromyalgia. The number of tender points where pain is reported is recorded
Average Pain Threshold | At baseline, then at the 2, 4 and 8 week visits
  Patients are examined for pain at the 18 characteristic tender points. The results of all the sites are added and divided by 18 to give an average pain threshold
Fibromyalgia Impact Questionaire | At baseline, then again at weeks 2, 4 and 8.
  Self-administered questionnaire that evaluates physical function, work status, depression anxiety, sleep, pain, stiffness, fatigue and well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Galimova, MD, Principal Investigator — The Royal College of Physicians and Surgeons of Canada; Ryan Skrabek, MD, Study Chair — University of Manitoba
Locations (1):
- Rehabilitation Hospital, Winnipeg, Manitoba, Canada